CLINICAL TRIAL: NCT00189111
Title: Non-invasive Cardiac Screening in High Risk Patients -The GROUND Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clinical Research Office Imaging Division (Other)
Responsible Party: Sponsor-Investigator, Clinical Research Office Imaging Division, Clinical research coordinator, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: METC.2004.100-GROUND
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2016-11

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease; computed tomography; cardiac asymptomatic; dobutamine magnetic resonance imaging
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Therapeutics

INTERVENTIONS:
Procedure: Cardiac Imaging + Treatment

SUMMARY:
The purpose of this study is to find out if subjecting cardiac high risk patients to non invasive cardiac imaging, followed by treatment will improve survival and quality of life

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is a common disease associated with a considerably increased risk of future events and with a high prevalence of coronary artery disease (CAD). Improvement of the prognosis of this patient group is needed. Screening for CAD has become an option with recent developments in CT-angiography and MR stress testing. It is unknown if high-risk patient groups benefit from screening through non-invasive cardiac imaging. Therefore we propose to study whether a cardiac imaging algorithm, using non-invasive imaging techniques followed by evidence-based treatment will reduce the risk of cardiovascular disease in cardiac asymptomatic PAD patients.

The GROUND study is designed as a prospective, multi-center, randomized clinical trial. Patients with peripheral arterial disease, but yet without a history of symptomatic cardiac disease will be asked to participate. All patients receive a proper therapeutic advice before randomization. Half of the recruited patients will enter the 'control group' and only receive CT calcium scoring. The other half of the recruited patients (index group) will undergo the non invasive cardiac imaging algorithm followed by evidence-based treatment. First patients undergo CT calcium scoring and CT angiography. Patients with a left main (or equivalent) coronary artery stenosis on CT angiography will be referred to a cardiologist without further imaging. All other patients in this group will undergo Dobutamine Stress Magnetic Resonance (DSMR) testing. Patients with a DSMR positive for ischemia will also be referred to a cardiologist. Most referred patients will very likely undergo conventional coronary artery angiography and cardiac interventions (CABG or PCI) if indicated. All participants of the trial will enter a 5 year follow up period for the occurrence of future cardiovascular events. Interim analysis will take place and based on power calculations about 1200 patients are needed to reach significance.

Implications The GROUND study will provide new insight into the question whether non-invasive cardiac imaging reduces the risk of cardiovascular events in patients with peripheral arterial disease, but yet without symptoms of coronary artery disease as an example of a high risk patient group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peripheral arterial disease, diagnosed by the vascular surgeon
* Patients must provide consent in writing after proper education and discussion with the treating physician and/or research physician
* Patients must be aged 50 years or over

Exclusion Criteria:

* History of symptomatic cardiac disease
* Cardiac rhythm other than sinus
* Unable to sustain a breath-hold for 25 seconds
* Asthma (contraindication beta-blockers)
* Contra-indications to MRI examination.
* Contra-indications to iodine contrast.
* Severe arterial hypertension (>220/120 mmHg)
* Significant aortic stenosis
* Unable to remain in supine position for at least 60 minutes
* Morbidly obese (BMI > 40)
* Renal insufficiency (creatinine >140mmol/l)
* Severe physical deterioration due to concomitant illness
* Language barrier
* Acute coronary syndrome
* Contra-indications to dobutamine

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2005-01; Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
cardiovascular mortality
cardiovascular morbidity

SECONDARY OUTCOMES:
Fatal and non-fatal myocardial infarction
Fatal and non-fatal stroke
Vascular interventions
Amputation
Aortic rupture
End stage renal failure
Extra cranial hemorrhage
Complications of CABG or PTCA
All cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: W. Mali, PhD, Principal Investigator — UMC Utrecht; M. Oudkerk, PhD, Principal Investigator — University Medical Center Groningen; M.L. Bots, PhD, Principal Investigator — Julius Center, University Medical Center Utrecht; F. Zijlstra, PhD, Principal Investigator — University Medical Center Groningen
Locations (5):
- Netherlands (5):
  - Bronovo Hospital, The Hague, South Holland
  - Meander Medical Center, Amersfoort, Utrecht
  - St. Antonius Hospital, Nieuwegein, Utrecht
  - University Medical Center Groningen, Groningen
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] de Vos AM, Rutten A, van de Zaag-Loonen HJ, Bots ML, Dikkers R, Buiskool RA, Mali WP, Lubbers DD, Mosterd A, Prokop M, Rensing BJ, Cramer MJ, van Es HW, Moll FL, van de Pavoordt ED, Doevendans PA, Velthuis BK, Mackaay AJ, Zijlstra F, Oudkerk M. Non-invasive cardiac assessment in high risk patients (The GROUND study): rationale, objectives and design of a multi-center randomized controlled clinical trial. Trials. 2008 Aug 1;9:49. doi: 10.1186/1745-6215-9-49. PMID 18673542